CLINICAL TRIAL: NCT02709096
Title: BPX-01 Minocycline 1% Topical Gel for Reduction of Propionibacterium Acnes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioPharmX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPX-01-C02
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BPX-01, 1% Topical Gel (Experimental): BPX-01, 1% Topical Gel; applied once daily to the face for four weeks.
  Interventions: Drug: BPX-01, 1% Topical Gel
- BPX-01, Vehicle Gel (Placebo Comparator): BPX-01, Vehicle Gel; applied once daily to the face for four weeks.
  Interventions: Drug: BPX-01 Vehicle Gel

INTERVENTIONS:
Drug: BPX-01, 1% Topical Gel — topical gel, applied to the forehead, cheeks, nose and chin
  Other Names: BPX-01 Topical Gel
  Arms: BPX-01, 1% Topical Gel
Drug: BPX-01 Vehicle Gel — topical gel, applied to the forehead, cheeks, nose and chin
  Other Names: BPX-01 Vehicle
  Arms: BPX-01, Vehicle Gel

SUMMARY:
This is a Phase 2a study which is being conducted in healthy volunteers in order to evaluate the comparative reduction of Propionibacterium acnes in-vivo following once daily topical administration of BPX-01 Minocycline 1% Topical Gel (BPX-01) or BPX-01 Vehicle control.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the comparative reduction of Propionibacterium acnes (P. acnes) in-vivo following once daily topical administration of BPX-01 Minocycline 1% Topical Gel or BPX-01 Vehicle control Gel.

A secondary objective is to assess the tolerance of the treatment regimen versus a vehicle control. Safety laboratory data (chemistry and hematology) and plasma levels of minocycline are also of significant interest to the sponsor.

This is a single center, randomized, double blind, two-cell, vehicle controlled P. acnes study. All subjects will be randomized 2:1 to 1% BPX-01 or vehicle control to be applied as a topical gel once daily for four (4) weeks.

This is a six (6) week study with a four (4) week treatment period and a two (2) week post treatment follow up visit. The clinical endpoint is in-vivo quantification of P.acnes. The safety/tolerance endpoints are; observer reported: erythema, scaling-peeling, edema, and subject reported: tightness, burning-stinging, and itching. Plasma levels of minocycline and basic hematology and chemistry laboratory values will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy, adult male and/or female volunteer 18 to 40 years of age with no past or present history of any significant disease based on PI discretion;
2. If female, must be post-menopausal, surgically sterile, or using effective birth control methods with a negative urine pregnancy test at the Screening and Baseline visits (female subjects of childbearing potential only);
3. Show a high degree of fluorescence of the face under a Wood's lamp at the screening visit.
4. Be willing to refrain from using antimicrobial topical products for the duration of study participation;
5. Be willing to return to the study center for all study visits;
6. Be willing to follow all study instructions and adhere to study restrictions;
7. Provide informed consent to the study procedures and restrictions

Exclusion Criteria:

1. Have a history of skin disease or presence of skin condition the PI believes would interfere with the study;
2. Females who report that they are pregnant, planning a pregnancy or breastfeeding or those females who are of child bearing potential, that test positive with a urine pregnancy test;
3. Have conditions or factors that the PI believes may affect the response of the skin or the interpretation of the results;
4. Participated in any clinical study within the previous 30 days, be concurrently participating in other studies, or be involved in any aspect of test administration;
5. Use of topical or systemic antibiotics or other products within the previous 4 weeks prior to baseline, that influence P. acnes counts;
6. Are known to be allergic to any of the test product(s) or any components in the test product(s);
7. Have a history of significant medical condition/disease that the PI believes may affect the response of the skin or the interpretation of the results;
8. Has any other condition that, in the opinion of the Investigator or his designee, could interfere with the subject's ability to use the treatment as instructed, alter their treatment response, or affect their ability to complete the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lessin, MD, Principal Investigator — KGL, Inc.
Locations (1):
- KGL Skin Study Center, Broomall, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BPX-01, 1% Topical Gel | BPX-01, Vehicle Gel
Started | 22 | 11
Completed | 21 | 10
Not Completed | 1 | 1
Not completed — non-compliance | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BPX-01, 1% Topical Gel | BPX-01, Vehicle Gel | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Continuous [Mean (Full Range); unit: years] | 32 [19 to 41] | 34 [24 to 40] | 32 [19 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 20 | 9 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Logarithmic Change in Colony Counts of Facial Propionibacterium Acnes
Description: P. Acnes cultures will be collected using the modified Kligman Method at each study visit. After plating, the samples will be cultured for 7 days and then evaluated.
Time Frame: Cultures will be evaluated at Baseline, Week 1, Week 2, Week 4 and Week 6. Values reported at week 4 compared to baseline.
Population: Per protocol population included all subjects with evaluable data and no major protocol violations.
Measure: Mean (Standard Deviation); unit: log change in colony forming units
Arm/Group | BPX-01, 1% Topical Gel | BPX-01, Vehicle Gel
Number analyzed (Participants) | 17 | 7
log change in colony forming units | -1.0376 (0.5479) | -0.4614 (0.4042)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | BPX-01, 1% Topical Gel | BPX-01, Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/11
Other Adverse Events (participants affected / at risk) | 4/22 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPX-01, 1% Topical Gel (N=22) | BPX-01, Vehicle Gel (N=11)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPX-01, 1% Topical Gel (N=22) | BPX-01, Vehicle Gel (N=11)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No